CLINICAL TRIAL: NCT03609437
Title: Impaired Endothelial Glycocalyx Integrity and Arterial Elastic Properties in Patients With Embolic Stroke of Undetermined Source (ESUS)
Brief Title: Impaired Endothelial Integrity in Patients With Embolic Stroke of Undetermined Source (ESUS)
Acronym: ESUS
Status: Active, not recruiting | Type: Observational
Sponsor: University of Athens (Other)
Responsible Party: Principal Investigator, Ignatios Ikonomidis, Dr Ignatios Ikonomidis,MD,PhD,FESC Associate Professor, University of Athens
Other Study IDs: esus-endothelium-attikon
Record Dates: First submitted 2018-07-15; First posted 2018-08-01 (Actual); Last update posted 2025-07-15 (Actual); Status verified 2025-07

CONDITIONS: Embolic Stroke of Undetermined Source; Endothelial Dysfunction
Keywords: Embolic stroke; Arterial stiffness; Endothelial function; Endothelial glycocalyx; Left ventricular function; Oxidative stress
MeSH Terms: conditions — Embolic Stroke

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Plasma
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (5):
- ESUS patients: Acute ischemic stroke patients satisfying embolic stroke of undetermined source (ESUS) diagnostic criteria.
- Controls: Healthy volunteers (colleagues, friends, relatives and others).
- Lacunar stroke patients: Acute ischemic stroke patients satisfying lacunar stroke diagnostic criteria
- Cardioembolic stroke patients: Acute ischemic stroke patients satisfying cardioembolic stroke diagnostic criteria
- Atherosclerotic stroke patients: Acute ischemic stroke patients satisfying atherosclerotic stroke diagnostic criteria

SUMMARY:
The investigators will measure endothelial glycocalyx, aortic elastic properties, oxidative stress, and their association with left ventricular (LV) and left atrial (LA) function in ESUS, cardioembolic, atherosclerotic, lacunar strokes and age- and sex-adjusted healthy individuals.

DETAILED DESCRIPTION:
Investigators plan to include male and female patients, aged 18 to 75 years old admitted and hospitalized in the 2nd Neurology Department of Attikon University Hospital for Acute Ischemic Stroke, based on the Trial of Org 10172 in Acute Stroke Treatment TOAST classification. The TOAST classification consists of five categories: 1) large artery atherosclerosis (atherothrombotic), 2) cardioembolic, 3) small artery occlusion (lacunar), 4) stroke of undetermined etiology (ESUS).

In participants (patients and controls) the investigators plan to measure and compare: a) perfused boundary region (PBR) of the sublingual arterial microvessels (range 5-25 micrometers), a marker inversely related with glycocalyx thickness, b) pulse wave velocity (PWV), central systolic blood pressure (cSBP) and augmentation index (AIx), c) LV Global Longitudinal strain (GLS), d) LA volume and strain using speckle-tracking strain imaging, e) Malondialdehyde (MDA), as an oxidative stress marker.

ELIGIBILITY:
Inclusion Criteria:

The investigators plan to include participants with Acute Ischemic Stroke, based on the TOAST classification : 1) large artery atherosclerosis (atherothrombotic), 2) cardioembolic, 3) small artery occlusion (lacunar), 4) stroke of undetermined etiology (ESUS). According to the TOAST classification, diagnoses are based on clinical presentation and on data collected by exams such as brain imaging (CT/MRI), cardiac imaging (echocardiography) and laboratory tests for the prothrombotic state. The diagnosis of Embolic Stroke of Undetermined Source (ESUS) was established based on the criteria defined by the Cryptogenic Stroke/ESUS International Working Group.

Exclusion Criteria

1. presence of acute haemorrhagic stroke,
2. the presence of stroke of other determined etiology,
3. the history of previous Ischemic stroke and/or Myocardial Infarction (MI),
4. hypercoagulable state,
5. active malignancy
6. severe chronic kidney disease (eGFR<30 ml/minute). These exclusion criteria are applied to both patients and control subjects.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The study population will consist of 172 consecutive patients with Ischemic stroke of undetermined source (ESUS) that fulfill inclusion criteria and 43 healthy volunteers of similar age and sex (control group)
Sampling Method: Non-Probability Sample
Enrollment: 215 (Estimated)
Dates: Start 2018-01-01 (Actual); Primary Completion 2025-10-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Comparison of endothelial glycocalyx thickness between patients with embolic stroke of undetermined source (ESUS), cardioembolic, atherosclerotic, lacunar strokes and controls | Baseline
  Investigators will assess endothelial glycocalyx thickness by evaluating perfused boundary region (PBR, micrometers) of the sublingual arterial microvessels (range 5-25 micrometers) for patients with embolic stroke of undetermined source (ESUS), cardioembolic, atherosclerotic, lacunar strokes and controls.

SECONDARY OUTCOMES:
Comparison of arterial stiffness between patients with embolic stroke of undetermined source (ESUS), cardioembolic, atherosclerotic, lacunar strokes and controls. | Baseline
  Investigators aim to evaluate arterial stiffness by pulse wave velocity (PWV,m/sec) using tonometry in patients with embolic stroke of undetermined source (ESUS), cardioembolic, atherosclerotic, lacunar strokes and controls.
Assessment of left ventricular performance in patients with embolic stroke of undetermined source (ESUS), cardioembolic, atherosclerotic, lacunar strokes and controls. | Baseline
  Investigators plan to assess left ventricular global longitudinal strain (GLS, %) in patients with embolic stroke of undetermined source (ESUS), cardioembolic, atherosclerotic, lacunar strokes and controls.
Serum malondialdehyde levels in patients with embolic stroke of undetermined source (ESUS), cardioembolic, atherosclerotic, lacunar strokes and controls. | Baseline
  Investigators plan to compare serum malondialdehyde levels in patients with embolic stroke of undetermined source (ESUS) and controls.
Assessment of left atrial performance in patients with embolic stroke of undetermined source (ESUS), cardioembolic, atherosclerotic, lacunar strokes and controls. | Baseline
  Investigators plan to compare left atrial strain (LA strain) in patients with embolic stroke of undetermined source (ESUS), cardioembolic, atherosclerotic, lacunar strokes and controls.

CONTACTS AND LOCATIONS:
Overall Officials: Ignatios Ikonomidis, Principal Investigator — University of Athens
Locations (1):
- Konstantinos Katogiannis, Athens, Attica, Greece

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Ikonomidis I, Frogoudaki A, Vrettou AR, Andreou I, Palaiodimou L, Katogiannis K, Liantinioti C, Vlastos D, Zervas P, Varoudi M, Lambadiari V, Triantafyllidi H, Pavlidis G, Efentakis P, Tsoumani M, Tsantes AE, Parissis J, Revela I, Andreadou I, Tsivgoulis G. Impaired Arterial Elastic Properties and Endothelial Glycocalyx in Patients with Embolic Stroke of Undetermined Source. Thromb Haemost. 2019 Nov;119(11):1860-1868. doi: 10.1055/s-0039-1694752. Epub 2019 Aug 17. PMID 31421641